CLINICAL TRIAL: NCT03610100
Title: A Phase III, Open Label, Multicentre Randomised Clinical Study Comparing Acelarin (NUC-1031) With Gemcitabine in Patients With Metastatic Pancreatic Carcinoma
Brief Title: Acelarin First Line Randomised Pancreatic Study
Acronym: ACELARATE
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Suspended to recruitment following TSC review on efficacy and toxicities
Sponsor: The Clatterbridge Cancer Centre NHS Foundation Trust (Other)
Collaborators: Cancer Research UK (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISRCTN16765355
Record Dates: First submitted 2016-09-27; First posted 2018-08-01 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-05

CONDITIONS: Pancreatic Acinar Carcinoma; Pancreatic Neoplasms
Keywords: Pancreatic; Neoplasms; Metastatic; Gemcitabine; Gemzar; Phosphoramidate; Cytidine Aminohydrolase; Deoxycytidine Kinase; Nucleoside Transport Proteins; hENT1 protein, human
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — NUC-1031; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acelarin (NUC-1031) (Experimental): 825 mg/m2 administered intravenously over 15 to 30 minutes on days 1, 8 and 15 of a 28 day cycle.
  Patients will be seen on a weekly basis during the time they are on active treatment and will be treated until disease progression.
  Interventions: Drug: Acelarin
- Gemcitabine (Active Comparator): Gemcitabine: 1000mg/m2 administered intravenously as a 30 minute infusion on days 1, 8 and 15 of a 28 day cycle.
  Patients will be seen on a weekly basis during the time they are on active treatment and will be treated until disease progression.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Acelarin — 825 mg/m2 administered intravenously over 15 to 30 minutes on days 1, 8 and 15 of a 28 day cycle. Number of Cycles: until disease progression or unacceptable toxicity develops.
  Other Names: NUC-1031
  Arms: Acelarin (NUC-1031)
Drug: Gemcitabine — 1000 mg/m2 administered intravenously as a 30 minute infusion on days 1, 8 and 15 of a 28 day cycle. Number of Cycles: until disease progression or unacceptable toxicity develops.
  Other Names: Gemzar
  Arms: Gemcitabine

SUMMARY:
The primary purpose of this study is to assess whether Acelarin (NUC-1031) is superior to gemcitabine in terms of overall survival for treatment of patients with metastatic pancreatic carcinoma. In addition disease progression, quality of life and comparative safety will be evaluated. Secondary objectives are to compare between the two treatment groups the following:

* Progression Free Survival (PFS)
* Radiological Response and disease control rate
* Toxicity and safety
* Quality of Life

Additional, exploratory objectives are to discover and validate possible biomarkers to predict additional benefit of Acelarin (NUC-1031) over gemcitabine alone.

DETAILED DESCRIPTION:
Pancreatic cancer remains the most lethal of solid tumours with little progress being made to improve patient outcomes over the past 30 years of research. The incidence in the UK is approximately 9,000 new cases per year and, with a 5 year survival remaining at just 3%, mortality approximates incidence. These dismal outcomes reflect:

1. Advanced stage at presentation such that only a minority of patients are suitable for surgery with curative intent;
2. High rates of recurrence even in those undergoing radical surgery;
3. Limited efficacy of systemic therapies.

   Until recently, the mainstay of systemic therapy for advanced pancreatic cancer was gemcitabine, based on the pivotal study in 1997 by Burris et al., reporting a survival and clinical benefit when compared with 5-FU. However, this benefit is modest with median and 1-year survival of approximately 6 months and 20% respectively for patients with metastatic disease. Combination chemotherapy has shown more promising results but at the expense of significant toxicity limiting this to younger patients with good performance status.

   Although these chemotherapy combinations confer a survival advantage over gemcitabine, their use is restricted to a cohort of patients able, and willing, to tolerate additional toxicity. Pancreatic cancer is commonly associated with:

   (i) increasing age; (ii) co-morbidities (for example, diabetes mellitus which, if associated with peripheral neuropathy, may limit the safe administration of neurotoxic drugs such as oxaliplatin and nab-paclitaxel); (iii) symptoms that negatively impact on performance status; (iv) biliary obstruction requiring stenting, with associated risks of sepsis and impaired drug metabolism.

   Thus, for a large proportion of patients single agent gemcitabine remains an appropriate standard chemotherapy. For this group of patients, more efficacious and better tolerated treatment is required.

   The study is being performed to investigate whether Acelarin provides improvement in overall survival compared with gemcitabine. This is a pivotal study in this indication and will represent the landmark data for whether there is additional benefit from Acelarin in pancreatic cancer.

   Gemcitabine monotherapy, the control arm, remains a standard of care in this disease. The only treatments that have shown improved outcome over gemcitabine are Folfirinox and nab-paclitaxel in combination with gemcitabine. However, the application of these regimens to a large proportion of patients with pancreatic cancer is limited by the potential for significant toxicities.

   Acelarin (NUC-1031) is a first-in-class nucleotide analogue, which uses novel phosphoramidate technology to overcome the key cancer resistance mechanisms associated with gemcitabine.

   Acelarin is synthesised as a pre-activated molecule bearing one protected phosphate group, termed the phosphoramidate motif, imparting several potential advantages to this new agent over gemcitabine:
   * Acelarin (NUC-1031) overcomes the reliance on nucleoside transporters to cross the cellular membrane for effective uptake by the cancer cells.
   * Acelarin (NUC-1031) presents the cell with an already partially activated (monophosphate) form of the nucleoside, thereby obviating the need for the rate limiting initial kinase activation.
   * Acelarin (NUC-1031) is protected from enzymatic breakdown (especially by deaminases and phosphorylases) resulting in greater stability and a reduction in the generation of toxic metabolites.

   The clinical relevance of these resistance mechanisms has been well documented.

   Multiple active nucleoside transporters located in the cell membrane carry out the transport of nucleoside analogues, such as gemcitabine, into the cells. The human equilibrative nucleoside transporter, hENT1 mediates the majority of gemcitabine uptake. It is therefore expected that hENT1-deficient cells are highly resistant to gemcitabine (Achiwa et al., Cancer Sci. 2004).

   Nucleoside transport deficiency is an important predictive factor for gemcitabine response in patients with cancer. Spratlin et al.,demonstrated that the presence of nucleoside transporters correlated with improved response to gemcitabine and OS in patients with pancreatic cancer (Spratlin et al Clin Cancer Res. 2004). Patients expressing hENT1 had a median survival of 13 months compared to only 4 months in patients with little or no hENT1 activity.

   Acelarin has been shown to overcome the need for hENT1 active transport to enter the cancer cells. The greater lipophilicity allows Acelarin to cross the cell membrane independently of nucleoside transporters.

   To become active, nucleoside analogues require sequential steps of phosphorylation within the cancer cells. Deficiency in dCK is a frequently described form of in-vitro and in-vivo inherent as well as acquired resistance to gemcitabine. Acelarin is synthesised as a monophosphate agent and, as such, has by-passed the rate limiting step of kinase-dependent activation.

   Acelarin bears a phosphoramidate moiety on the ribose 5' carbon, which protects the compound from deamination (Slusarczyk et al J Med Chem 2014) , which may confer considerable survival advantages and a more favourable safety profile (Ghazali et al JCO 322:5s, 2014).

   It is planned to perform this study in approximately 40 UK centres with additional centres in Europe and the USA with a centre defined as the primary institution of the clinical investigator. Recruitment will be competitive and 328 patients will be randomised in a 1:1 fashion.

   Randomisation will be stratified by ECOG performance status (PS) (0/1 vs 2).

   Baseline radiographic assessment of disease will be performed within 28 days prior to first treatment and first treatment will be delivered within 8 days of randomisation or the earliest screening procedure, e.g. blood samples, CT scan whichever is sooner as follows:

   Arm A (experimental arm): Acelarin (NUC-1031)

   Acelarin: 825 mg/m2 administered intravenously over 15 to 30 minutes on days 1, 8 and 15 of a 28 day cycle

   Arm B (standard therapeutic arm): Gemcitabine

   Gemcitabine: 1000mg/m2 administered intravenously as a 30 minute infusion on days 1, 8 and 15 of a 28 day cycle

   Patients will be seen on a weekly basis during the time they are on active treatment and will be treated until disease progression. At the completion of therapy, an end-of therapy visit must be completed within 7 days after the decision is made to discontinue all therapy. This must be a full assessment consisting of physical exam, Performance Status, ECG, haematology and chemistry profile and toxicity/AE assessments, after which follow up will then occur every 12 weeks. CT scans of the chest, abdomen and pelvis will take place at screening then every 12 weeks thereafter until disease progression as per RECIST 1.1.

   No further anti-tumour treatment will be initiated until progression of disease. AE information will be collected until at least 30 days after the last dose of study therapy is administered or until all study therapy-related AEs have resolved, stabilised or been deemed irreversible and a 30 day safety follow up should be performed at this point.

   A phase I/II clinical study has established the RP2D and schedule for Acelarin as 825 mg/m2 administered intravenously on days 1, 8 and 15 of a 28 day cycle. Two dose limiting toxicities were observed (grade 3 transaminitis at 725mg/m2 and grade 4 thrombocytopenia at 750mg/m2). Otherwise treatment was well-tolerated with no unexpected adverse events. Adverse events were generally mild to moderate with the most common grade 1 and 2 AEs being anaemia, fatigue, transaminitis and thrombocytopenia. Only three patients experienced grade 4 AEs: thrombocytopenia, hypomagnesaemia and sepsis.

   The following precautionary measures will also be put in place:
   * Assessment of full blood count, renal function and liver function will be made prior to each administration of Acelarin.
   * The occurrence of haematological toxicity including neutropenia and thrombocytopenia which requires dose adjustment is specified in the protocol.
   * The effect of renal impairment on exposure to Acelarin in patients with renal impairment is not known. Therefore study entry is restricted to patients with creatinine clearance ≥ 30mL/minute.
   * Acelarin should not be administered to pregnant women. A negative pregnancy test should be confirmed before administration of Acelarin for all women of childbearing age.
   * There is no known antidote for Acelarin, and treatment of AEs associated with its use should be for the underlying adverse symptoms.
   * Since Acelarin will be reconstituted in specialist oncology pharmacies and administered by experienced chemotherapy-trained nurses via intravenous injection, overdose is considered to be highly unlikely. There is no specific treatment for an overdose of Acelarin. In case of overdose, therapy may be interrupted, and any adverse reactions treated symptomatically.

   Assessment of full blood count, renal function and liver function will be made prior to each administration of gemcitabine.

   The occurrence of haematological toxicity including neutropenia and thrombocytopenia which requires dose adjustment is specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically or cytologically proven pancreatic ductal adenocarcinoma or undifferentiated carcinoma of the pancreas.
* Metastatic disease precluding curative surgical resection or definitive locally directed therapies such as chemo radiation. Patients who have relapsed following previously resected pancreatic cancer can be included.
* Contrast enhanced computerised tomography (CT) scan of the thorax, abdomen and pelvis within 28 days prior to commencing treatment.
* Unidimensionally measurable disease.
* ECOG performance status 0, 1 or 2 where combination chemotherapy is not deemed appropriate or is declined by the patient.
* Platelets ≥100 x 109/l; WBC ≥ 3 x 109/l; neutrophils ≥ 1.5 x 109/l at entry.
* Documented life expectancy > 3 months.
* Informed written consent.

Exclusion Criteria:

* Laboratory results:

  * Serum bilirubin ≥ 1.5x the upper limit of reference range (ULRR).
  * Haemoglobin < 10G/dl.
  * Creatinine clearance < 30 mL/minute (calculated by Cockcroft-Gault formula).
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 x ULN or > 5x ULN if judged by the investigator to be related to liver metastases.
* Medical or psychiatric conditions compromising informed consent.
* Intracerebral metastases or meningeal carcinomatosis.
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardize compliance with the protocol.
* Pregnancy or breast feeding.
* Previous chemotherapy for locally advanced and metastatic disease. Adjuvant chemotherapy for resected pancreatic cancer will be permitted provided that chemotherapy was completed > 12 months previously.
* Radiotherapy within the last 4 weeks prior to start of study treatment.
* Concurrent malignancies or invasive cancers diagnosed within past 5 years except for adequately treated basal cell carcinoma of the skin, in situ carcinoma of the uterine cervix or resected pancreatic cancer.
* Hypersensitivity to gemcitabine or any of the excipients of gemcitabine or Acelarin (NUC-1031).
* All men or women of reproductive potential, unless using at least two contraceptive precautions, one of which must be from the list below, the other must be a condom* or abstaining from sexual intercourse, until six months after treatment has ended:

  * Combined (oestrogen and progesterone containing) hormonal contraception associated with inhibition of ovulation: either oral, intravaginal or transdermal.
  * Progesterone-only hormonal contraception associated with inhibition of ovulation: either oral, injectable or implantable.
  * Intra-uterine device (IUD)
  * Intra-uterine hormone-releasing system (IUS)
  * Bilateral tubal occlusion
  * Vasectomised partner *Male or female condom with or without spermicide is not an acceptable method of contraception alone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2015-12; Primary Completion 2020-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants that have survived throughout treatment and also into follow-up, as measured by the primary cause of death and date of death CRFs. | 4 years

SECONDARY OUTCOMES:
Number of participants that survive progression-free and for how long, as assessed by 12-weekly CT scan assessments per RECIST v1.1 and end of study CRF to capture the reasons for coming off study. | 4 years
Number of participants that show an objective response, as demonstrated by 12-weekly CT scan assessments per RECIST v1.1. | 4 years
Number of participants deemed to have disease control, as demonstrated by 12-weekly CT scan assessments per RECIST v1.1. | 4 years
Number of patients with treatment-related adverse events as assessed by CTCAE v4.03. Toxicity is assessed by CTCAE v4.03 alongside Quality of Life Questionnaires, QLQ-C30 and QLQ-PAN26. | 4 years

OTHER OUTCOMES:
Discovery of possible biomarkers which may predict any additional benefit of Acelarin over gemcitabine. These will be assessed from plasma, cell pellet and serum samples collected from participants throughout the trial. | 4 years
  To validate candidate predictive biomarkers, baseline patient samples will be analysed by Luminex technology. Paraffin embedded formalin fixed pancreatic cancer biopsy tissue samples will be used for analysis of candidate predictive biomarkers. Transcripts that will be assayed with RNAScope and scored for staining are: hENT1; CDA, dCK; RRM1 & RRM2. RNAscope will be used to detect mRNA expression by using a site directed probe, to a particular sequence in the gene of interest, which is then amplified and stained. This enables quantification of the mRNA expression and allows subsequent survival analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Palmer, BSC, PhD, Principal Investigator — University of Liverpool
Locations (1):
- Cancer Research UK Liverpool Cancer Trials Unit, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Von Hoff DD, Ervin TJ, Arena FP, et al: "Randomized phase III study of weekly nab-paclitaxel plus gemcitabine versus gemcitabine alone in patients with metastatic adenocarcinoma of the pancreas (MPACT)". 2013 Gastrointestinal Cancers Symposium. J Clin Oncol 31, 2013 (suppl 4; abstract: LBA148)
- [Background] Ghazaly, E.A. et al. "ProGem1: Phase I first-in-human study of the novel nucleotide NUC-1031 in adult patients with advanced solid tumors" J Clin Oncol 31, 2013 (suppl; abstr 2576)
- [Background] de Sousa Cavalcante L, Monteiro G. Gemcitabine: metabolism and molecular mechanisms of action, sensitivity and chemoresistance in pancreatic cancer. Eur J Pharmacol. 2014 Oct 15;741:8-16. doi: 10.1016/j.ejphar.2014.07.041. Epub 2014 Jul 30. PMID 25084222
- [Background] Achiwa H, Oguri T, Sato S, Maeda H, Niimi T, Ueda R. Determinants of sensitivity and resistance to gemcitabine: the roles of human equilibrative nucleoside transporter 1 and deoxycytidine kinase in non-small cell lung cancer. Cancer Sci. 2004 Sep;95(9):753-7. doi: 10.1111/j.1349-7006.2004.tb03257.x. PMID 15471562
- [Background] Spratlin J, Sangha R, Glubrecht D, Dabbagh L, Young JD, Dumontet C, Cass C, Lai R, Mackey JR. The absence of human equilibrative nucleoside transporter 1 is associated with reduced survival in patients with gemcitabine-treated pancreas adenocarcinoma. Clin Cancer Res. 2004 Oct 15;10(20):6956-61. doi: 10.1158/1078-0432.CCR-04-0224. PMID 15501974
- [Background] Ghazaly, E.A. et al. "ProGem1: A phase I/II study of a first-in-class nucleotide, Acelarin, in patients with advanced solid tumors" J Clin Oncol 32:5s, 2014 (suppl; abstr 2531)
- [Background] Sebastiani V, Ricci F, Rubio-Viqueira B, Kulesza P, Yeo CJ, Hidalgo M, Klein A, Laheru D, Iacobuzio-Donahue CA. Immunohistochemical and genetic evaluation of deoxycytidine kinase in pancreatic cancer: relationship to molecular mechanisms of gemcitabine resistance and survival. Clin Cancer Res. 2006 Apr 15;12(8):2492-7. doi: 10.1158/1078-0432.CCR-05-2655. PMID 16638857
- [Background] Kroep JR, van Moorsel CJ, Veerman G, Voorn DA, Schultz RM, Worzalla JF, Tanzer LR, Merriman RL, Pinedo HM, Peters GJ. Role of deoxycytidine kinase (dCK), thymidine kinase 2 (TK2), and deoxycytidine deaminase (dCDA) in the antitumor activity of gemcitabine (dFdC). Adv Exp Med Biol. 1998;431:657-60. doi: 10.1007/978-1-4615-5381-6_127. No abstract available. PMID 9598147
- [Background] Philip PA, Chansky K, LeBlanc M, Rubinstein L, Seymour L, Ivy SP, Alberts SR, Catalano PJ, Crowley J. Historical controls for metastatic pancreatic cancer: benchmarks for planning and analyzing single-arm phase II trials. Clin Cancer Res. 2014 Aug 15;20(16):4176-85. doi: 10.1158/1078-0432.CCR-13-2024. Epub 2014 Jun 9. PMID 24914040
- [Background] Slusarczyk M, Lopez MH, Balzarini J, Mason M, Jiang WG, Blagden S, Thompson E, Ghazaly E, McGuigan C. Application of ProTide technology to gemcitabine: a successful approach to overcome the key cancer resistance mechanisms leads to a new agent (NUC-1031) in clinical development. J Med Chem. 2014 Feb 27;57(4):1531-42. doi: 10.1021/jm401853a. Epub 2014 Feb 14. PMID 24471998
- [Background] Moore MJ, Goldstein D, Hamm J, Figer A, Hecht JR, Gallinger S, Au HJ, Murawa P, Walde D, Wolff RA, Campos D, Lim R, Ding K, Clark G, Voskoglou-Nomikos T, Ptasynski M, Parulekar W; National Cancer Institute of Canada Clinical Trials Group. Erlotinib plus gemcitabine compared with gemcitabine alone in patients with advanced pancreatic cancer: a phase III trial of the National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 2007 May 20;25(15):1960-6. doi: 10.1200/JCO.2006.07.9525. Epub 2007 Apr 23. PMID 17452677